CLINICAL TRIAL: NCT03778567
Title: The Effect of Telbivudine on Renal Function in Chronic Hepatitis B Patients With Mild to Moderate Renal Impairment
Brief Title: Renoprotective Effects of Telbivudine in Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Yuen Man Fung, Deputy Head of Department, The University of Hong Kong
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HKUCTR - 1639
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Hepatitis B, Chronic; Chronic Kidney Diseases
Keywords: chronic hepatitis B infection; telbivudine; chronic kidney disease; nucleotide analogue
MeSH Terms: conditions — Hepatitis B, Chronic; Renal Insufficiency, Chronic | interventions — Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lamivudine + nucleotide analogue (Other): At the time of recruitment (0 month, baseline), lamivudine is switched to telbivudine while adefovir or tenofovir disoproxil fumarate was continued
  Interventions: Drug: Telbivudine

INTERVENTIONS:
Drug: Telbivudine — CHB patients who are receiving adefovir or tenofovir disoproxil fumarate are recruited. At the time of recruitment (0 month, baseline), lamivudine is switched to telbivudine while adefovir or tenofovir disoproxil fumarate was continued. The patients are followed-up for 24 months.
  Other Names: lamivudine is switched to telbivudine

SUMMARY:
Renal impairment is common in patients with chronic hepatitis B infection. For those taking nucleotide analogues, renal toxicity of adefovir disoproxil (ADV) and tenofovir disoproxil fumarate (TDF) is a significant concern in chronic hepatitis B (CHB) patients. Early observational clinical data suggested that telbivudine (LdT) might have renoprotective effects. In this prospective study, consecutive CHB patients on combined lamivudine (LAM)+ADV/TDF are switched to LdT+ADV/TDF at recruitment and are followed up for 24 months. Estimated glomerular filtration rate (eGFR) is calculated with the Modification of Diet in Renal Disease (MDRD) equation. The effects of LdT on cell viability and expression of kidney injury or apoptotic biomarkers are investigated in cultured renal tubular epithelial cell line HK-2.

DETAILED DESCRIPTION:
Background

Both CHB and chronic kidney disease are major health issue affecting millions of persons worldwide. Based on a large European multicenter database, the Virgil-database, it is estimated that 15% and 4% of the CHB patients in Europe had mild (GFR 50-80ml/min) and moderate (GFR <50ml/min) renal impairment respectively . These group of patients require special attention as the nucleos(t)ides agents (NA) used in the treatment of CHB are cleared by kidneys and may worsen the kidney function. Recently, a subgroup analysis of the GLOBE study and 4 small prospective studies provide circumstantial evidence on the use of telbivudine (LDT) that can improve renal function in CHB patients. However, there are no prospective, controlled trials to date to evaluate the relationship between LDT and renal function.

Research plan and methodology

This is a prospective study in CHB patients treated with NA and pre-existing mild to moderate renal impairment defined as estimated GFR (eGFR) 30-90ml/min.

Aims

To compare the renal function of patients before and after switching lamivudine to telbivudine.

To determine any adverse events from switching other NA to telbivudine To determine any biochemical and virological change from switching other NA to telbivudine by checking ALT, HBV DNA at baseline, and at weeks 12, 24, 36, 48, 60, 72, 84, 96 and 108 weeks To determine any change in 24 hour urinary protein and urinary glucose level To determine the in vitro effects of telbivudine on renal tubular cells

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 70 years
2. Documented HBsAg positivity for at least 6 months. Patients can be either HBeAg positive AND HBV DNA < 9 log10 copies/mL or HBeAg negative AND HBV DNA < 7 log10 copies/mL
3. On combination therapy (lamivudine and tenofovir or lamivudine and adefovir) for at least 1 year
4. Documented serum creatinine at least in 2 separate occasions in the last 1 year before recruitment
5. MDRD eGFR 30-89ml/min at baseline

Exclusion Criteria:

1. Concomitant liver disease including chronic hepatitis C and/or D infection, Wilson's disease, autoimmune hepatitis, primary biliary cirrhosis and primary sclerosing cholangitis
2. Significant alcohol intake or drug abuse
3. Pregnant subjects
4. Patients with co-existing significant chronic kidney disease (e.g.post renal transplantation etc.)
5. Allergic to any of the medications involved in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-06-16 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Renal function change | 108 weeks
  Describe the change in renal function after 108 weeks of telbivudine switch

SECONDARY OUTCOMES:
Virologic suppression | 108 weeks
  Rate of virologic suppression
Adverse events | 108 weeks
  Rate of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Man-Fung Yuen, DSc, MD, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Mak LY, Liu SH, Yap DY, Seto WK, Wong DK, Fung J, Chan TM, Lai CL, Yuen MF. In Vitro and In Vivo Renoprotective Effects of Telbivudine in Chronic Hepatitis B Patients Receiving Nucleotide Analogue. Dig Dis Sci. 2019 Dec;64(12):3630-3641. doi: 10.1007/s10620-019-05717-0. Epub 2019 Jul 6. PMID 31280390